CLINICAL TRIAL: NCT02486471
Title: Is a Hemostatic Procedure Required After Biopsy of the Cervix Uteri in Women Undergoing Colposcopy for Cervical Dysplasia? A Multicenter Randomized Non-inferiority Trial
Brief Title: Hemostatic Procedure After Biopsy of the Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Responsible Party: Principal Investigator, Dr. med. Ziad Hilal, Dr. med. Ziad Hilal, Zydolab - Institute of Cytology and Immune Cytochemistry
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: COLPO-1
Record Dates: First submitted 2015-06-28; First posted 2015-07-01 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Uterine Cervical Dysplasia
Keywords: cervical dysplasia; colposcopy; haemostatic procedure; biopsy of the cervix uteri
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Vision, Ocular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observational approach (Other): Wait and see
  Interventions: Other: Wait and see
- Use of Monsel´s Paste (Active Comparator): cervical coagulation using a hemostatic agents, ie monsel´s paste
  Interventions: Procedure: Monsel´s Paste

INTERVENTIONS:
Procedure: Monsel´s Paste — surgical method to stop bleeding by using the hemostatic Agent monsel´s paste until no more bleeding is visible
  Arms: Use of Monsel´s Paste
Other: Wait and see — finishing examination without hemostatic intervention, awaiting spontaneous coagulation
  Arms: Observational approach

SUMMARY:
Cytological abnormalities of the Cervix uteri need to be clarified by colposcopy biopsy. To avoid bleeding after biopsy, monsel´s paste is a common used Agent. In a randomized clinical Trial the use of monsel´s paste after biopsy will be compared to no Intervention. The Primary outcome of the study is blood loss, secondary outcomes are pain, satisfaction of the patient and influence of Independent factors such as Age and Body mass index.

ELIGIBILITY:
Inclusion Criteria:

* abnormal pap smear
* first colposcopy ever

Exclusion Criteria:

* pregnancy
* bleeding disorder
* the use of blood thinner
* language barrier
* unwillingness to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Blood loss after 15 minutes (5-step visual analogue scale) | 15 minutes
  blood loss 15 minutes after biopsy will be measured judging the amount of blood on the sanitary napkin (5-step visual analogue scale)

SECONDARY OUTCOMES:
Blood loss after 3 hours (5-step visual analogue scale) | 3 hours
  blood loss 3 hours after biopsy will be measured judging the amount of blood on the sanitary napkin (5-step visual analogue scale)
Blood loss after 6 hours (5-step visual analogue scale) | 6 hours
  blood loss 6 hours after biopsy will be measured judging the amount of blood on the sanitary napkin (5-step visual analogue scale)
Blood loss after 24 hours (5-step visual analogue scale) | 24 hours
  blood loss 24 hours after biopsy will be measured judging the amount of blood on the sanitary napkin (5-step visual analogue scale)
Sensation of pain after 15 minutes (10-step visual analogue scale) | 15 minutes
  patients will score their pain Level using a 10-step visual analogue scale (VAS) 15 minutes after biopsy
Overall Sensation of pain after 24 hours (10-step visual analogue scale) | 24 hours
  patients will score their pain Level using a 10-step visual analogue scale (VAS) 24 hours after biopsy
Overall Satisfaction of the Patient after 24 hours (10-step visual analogue scale) | 24 hours
  patients will score their satisfaction Level using a 10-step visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, M. D., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (2):
- Germany (2):
  - Zydolab - Institute of Cytology and Immune Cytochemistry, Dortmund, North Rhine-Westphalia
  - Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No